CLINICAL TRIAL: NCT03796637
Title: Phase 2, Non-Interventional, Clinical Study to Assess Dystrophin Levels in Subjects With Nonsense Mutation Duchenne Muscular Dystrophy Who Have Been Treated With Ataluren for ≥9 Months
Brief Title: A Study to Assess Dystrophin Levels in Participants With Nonsense Mutation Duchenne Muscular Dystrophy (nmDMD) Who Have Been Treated With Ataluren
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTC124-GD-046-DMD; 2019-001691-11 (EudraCT Number)
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-02

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nmDMD Participants (Experimental): Participants who have been receiving ataluren, will be dosed daily 10 milligrams per kilogram (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening, for >=9 months from ongoing PTC-sponsored nmDMD clinical trials.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be administered as per the dose and schedule specified in the arm.
  Other Names: PTC124

SUMMARY:
This study is designed to generate additional data on the effect of ataluren for producing dystrophin protein in nonsense mutation nmDMD participants. This study will evaluate dystrophin levels from participants with nmDMD who currently have been receiving ataluren for ≥9 months.

The study will have a single visit (Visit 1).

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent/assent document(s) indicating that the participant (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial.
* Ambulatory (10 meters walk/run in less than [<] 30 seconds) and functional grade on the Brooke Upper Extremity Scale of a 1 or a 2.
* Currently being treated with ataluren 10, 10, 20 mg/kg for >=9 months, with no gap in treatment of greater than (>) 1 month, in an ongoing PTC-sponsored nmDMD clinical trial prior to study entry.
* Phenotypic evidence of duchenne muscular dystrophy (DMD) based on the onset of characteristic clinical symptoms or signs (for example, proximal muscle weakness, waddling gait, and Gowers' maneuver) by 6 years of age and an elevated serum creatine kinase (CK). Medical documentation of phenotypic evidence of DMD needs to be provided upon request by the medical monitor.
* Willing to undergo muscle biopsy.

Exclusion Criteria:

* Known contra-indication to muscle biopsy (such as bleeding or clotting disorders).
* Exposure to another investigational drug within 2 months prior to study enrollment or ongoing participation in any non-ataluren interventional clinical trial.
* Requirement for daytime ventilator assistance or any use of invasive mechanical ventilation via tracheostomy. Note: Evening non-invasive mechanical ventilation such as use of bilevel positive airway pressure (Bi-PAP) therapy is allowed.
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder), medical history, physical findings or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bibbiani, MD, Study Director — PTC Therapeutics, Inc.
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ataluren: Participants who had been receiving ataluren, were dosed daily 10 milligrams (mg)/kilogram (kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening, for ≥9 months from ongoing PTC-sponsored nmDMD clinical trials.
Period: Overall Study
Arm/Group | Ataluren
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants with a valid assessment of dystrophin level, as measured by electrochemiluminescence (ECL).
Groups:
- Ataluren: Participants who had been receiving ataluren, were dosed daily 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening, for ≥9 months from ongoing PTC-sponsored nmDMD clinical trials.
Arm/Group | Ataluren
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Dystrophin Levels as Measured by Electrochemiluminescence (ECL)
Description: The mean dystrophin protein levels were measured by ECL. Dystrophin levels are reported by muscle group (gastrocnemius, tibialis anterior, and across muscle locations). Results below the limit of quantitation were imputed as half of lower limit of quantitation (LLOQ). LLOQ = 0.5 micrograms (μg)/milliliter (mL)
Time Frame: Day 1 of biopsy
Population: ITT population included all enrolled participants with a valid assessment of dystrophin level, as measured by ECL.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mg
Arm/Group | Ataluren
Number analyzed (Participants) | 6
nanograms (ng)/mg
  Gastrocnemius | 0.0844 (0.05874)
  Tibialis Anterior | 0.1002 (0.08060)
  Across Muscle Locations | 0.1054 (0.08300)

2. Secondary Outcome: Dystrophin Protein Levels as Determined by Immunohistochemistry
Description: Dystrophin levels by IHC mean membrane stain density are reported by muscle group (gastrocnemius, tibialis anterior, and across muscle locations).
Time Frame: Day 1 of biopsy
Population: ITT population included all enrolled participants with a valid assessment of dystrophin level, as measured by ECL.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | Ataluren
Number analyzed (Participants) | 6
ng/mg
  Gastrocnemius | 0.28817 (0.220547)
  Tibialis Anterior | 0.26578 (0.226510)
  Across Muscle Locations | 0.30483 (0.218600)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Week 1
Description: Safety population included all participants who received at least 1 dose of ataluren.
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=6)
Puncture site discharge (General disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT03796637/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT03796637/SAP_001.pdf